CLINICAL TRIAL: NCT01678794
Title: Define in Humans With Compensated CHF and Renal Dysfunction, the Modulating Action of Chronic AT1 Receptor Blockade in Addition to ACE Inhibition on Cardiorenal and Humoral Function
Brief Title: CR Aim #2 - AT1 Receptor Blockade & ACE Inhibition Effect on Humoral Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Horng Chen, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-003284; 1R01HL084155-01A2 (NIH)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Cardiorenal Syndrome (CRS)
Keywords: Chronic heart failure (CHF); cardiac and renal dysfunction
MeSH Terms: conditions — Cardio-Renal Syndrome; Renal Insufficiency | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Candesartan (Experimental)
  Interventions: Drug: Candesartan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan — 4 mg once a day up to 13 day. dose will be doubled every 14-18 days as tolerated to a goal of 16 mg a day or highest dose tolerated
  Other Names: Atacand
  Arms: Candesartan
Drug: Placebo — 4 mg once a day up to 13 day. dose will be doubled every 14-18 days as tolerated to a goal of 16 mg a day or highest dose tolerated
  Arms: Placebo

SUMMARY:
To advance our understanding of the mechanisms of human cardiorenal syndrome with emphasis upon the interaction of diuretic therapy and the renal-angiotensin-aldosterone -system and cGMP pathway.

The belief is that the chronic AT1 receptor blockade in subjects with compensated CHF and renal dysfunction will improve renal function with increased sodium excretion, glomerular filtration rate and effective renal plasma flow and renal function reserve as compared to the response of placebo-treated subjects.

DETAILED DESCRIPTION:
IRB # 09-003284, "Specific Aims 2: Define in humans with compensated CHF and renal dysfunction, the modulating action of chronic AT1 receptor blockade in addition to ACE inhibition on cardiorenal and humoral function", involving 12 weeks of study drug (Candesartan or placebo) starting at 4 mg daily and doubling every 2 weeks to 16 mg, if tolerated. Safety labs are performed one week after each dose increase (end of weeks 1, 3 and 5), and in week 10 of the study. Participants are monitoring their blood pressure weekly, and are aware to watch for symptoms of hypotension (lightheadedness, dizziness, blurred vision). Renal clearance testing and ECHO are performed at the start and end of the 12 weeks of study medication in the 5-Domitilla Clinical Research Unit.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction of equal or less than 40% assessed by echocardiography, nuclear scan, MRI or left ventriculogram within the past 48 months.
* Stable New York Heart Association (NYHA) class II and III symptoms as defined by: no change in NYHA symptoms over the past 3 months, on stable doses of ACE inhibitor, beta blocker, digoxin and furosemide over the last 4 weeks and no episode of decompensated CHF over the past 6 months.
* Calculated creatinine clearance of equal or less than 80 ml/min and greater than 20 ml/min, using the MDRD formula assessed within the past 48 months and a confirmatory calculated creatinine clearance equal or less than 80 ml/min and greater than 20 ml/min at the time of enrollment.

Subjects who are already taking AT1 receptor blocker will be excluded. Aldosterone antagonist, antiarrhythmic medications and other vasodilators will be allowed; however, all medications must be at stable doses 4 weeks prior to enrollment. Subjects taking nonsteroidal anti-inflammatory drugs (NSAIDs) except aspirin will not be able to increase their medication dose for the duration of the study. Subjects will be excluded if they have had a prior diagnosis of intrinsic renal disease, including renal artery stenosis of > 50%, or if they meet any one of the exclusion criteria listed below.

Exclusion Criteria:

* Prior diagnosis of intrinsic renal diseases including renal artery stenosis of > 50%
* Peritoneal or hemodialysis within 90 days or anticipation that dialysis or ultrafiltration of any form will be required during the study period
* Hospitalization for decompensated CHF during the past 6 months
* Subjects that are taking AT1 receptor blockers
* Myocardial infarction within 6 months of screening
* Unstable angina within 6 months of screening, or any evidence of myocardial ischemia
* Significant valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* Severe congenital heart diseases
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* Second or third degree heart block without a permanent cardiac pacemaker
* Stroke within 3 months of screening, or other evidence of significantly compromised CNS perfusion
* ALT >1.5 times the upper limit of normal
* Serum sodium of < 125 mEq/dL or > 160 mEq/dL
* Serum potassium of < 3.5 mEq/dL or > 5.7 mEq/dL
* Serum digoxin level of > 2.0 ng/ml
* Hemoglobin < 9 gm/dl
* Other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data
* Received an investigational drug within 1 month prior to dosing
* Patients with an allergy to iodine.
* Female subject who is pregnant or breastfeeding
* In the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-02; Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Foundation
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Candesartan; Placebo: Subjects received 4 mg once a day up to 13 day. Dose was doubled every 14-18 days as tolerated to a goal of 16 mg a day or highest dose tolerated.
Period: Overall Study
Arm/Group | Candesartan | Placebo
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Candesartan | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (10.4) | 69.3 (14.2) | 68.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 17 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Glomerular Filtration Rate
Description: Glomerular Filtration Rate estimates how much blood passes through the glomeruli each minute. Glomeruli are the tiny filters in the kidneys that filter waste from the blood. Measured as ml/min/1.73 m2
Time Frame: baseline to 3 months
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73 m2
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 16 | 17
ml/min/1.73 m2 | -5 [-14.5 to 3.5] | 1.00 [-8.00 to 6.00]
Statistical Analysis 1: Comparison: Candesartan vs Placebo; Test type: Superiority; p = 0.26, t-test, 2 sided

2. Primary Outcome: Change in Urinary Sodium Excretion
Description: Urinary sodium excretion correlates with elevated blood pressure in subjects at low cardiovascular risk. The body continually monitors blood volume and sodium concentration. When either becomes too high, sensors in the heart, blood vessels, and kidneys detect the increases and stimulate the kidneys to increase sodium excretion, thus returning blood volume to normal. Measured as mEq/min
Time Frame: baseline to 3 months
Measure: Median (Inter-Quartile Range); unit: mEq/min
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 16 | 17
mEq/min | -8.50 [-30.50 to 48.50] | 10.00 [-53.00 to 66.00]
Statistical Analysis 1: Comparison: Candesartan vs Placebo; Test type: Superiority; p = 0.67, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 3 months.
Arm/Group | Candesartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 5/16 | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Candesartan (N=16) | Placebo (N=17)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased plasma creatinine (Investigations) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lightheadness (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT01678794/Prot_SAP_000.pdf